CLINICAL TRIAL: NCT00379652
Title: Community, Health Center, and Academic Medicine Partnership Project (CHAMPP)
Brief Title: Community Partnership to Examine Racial and Ethnic Differences in Health Care for Hypertension and Diabetes
Acronym: CHAMPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 410; R21HL083859-01 (NIH); 1R21HL083859-01 (NIH)
Record Dates: First submitted 2006-09-20; First posted 2006-09-22 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Hypertension; Diabetes Mellitis
Keywords: Community Health Centers; Diabetes; Blood Pressure, High
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Patient Education as Topic; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Active Comparator): Patient-based intervention
  Interventions: Behavioral: Patient Education and Support
- B (Active Comparator): Health center-based intervention
  Interventions: Behavioral: Medical Practice Improvement
- C (Active Comparator): Combination of patient and health center-based intervention
  Interventions: Other: Combination Intervention to Include Medical Practice Improvement and Patient Education and Support
- D (No Intervention): Control group: Neither patient-based nor center-based intervention

INTERVENTIONS:
Behavioral: Medical Practice Improvement — The details for the medical practice improvement intervention will be decided at a later date.
  Arms: B
Behavioral: Patient Education and Support — The details for the patient education and support intervention will be decided at a later date.
  Arms: A
Other: Combination Intervention to Include Medical Practice Improvement and Patient Education and Support — The details for this combination intervention will be decided at a later date.
  Arms: C

SUMMARY:
Hypertension and diabetes are among the most common chronic diseases in the United States. Racial and ethnic minority groups are more at risk for these diseases than the Caucasian population. This study will attempt to identify factors that contribute to racial and ethnic differences in hypertension and diabetes care among minority patients of community health centers (CHCs). This information will be used to design and implement programs to improve quality of care in these communities.

DETAILED DESCRIPTION:
Hypertension and diabetes are the primary contributors to today's high rates of heart disease and stroke, which are the first and third leading causes of death in the United States, respectively. African Americans and Hispanics have a higher risk of developing hypertension and diabetes than do Caucasians. They are also less likely to know that they have high blood pressure, are more prone to organ damage, and are more likely to die as a result of these chronic conditions. A significant number of African Americans and Hispanics are uninsured and receive care through publicly supported CHCs. It is important to identify factors that contribute to healthcare differences among the lower income, uninsured, and minority populations that are typically served by CHCs. In this study, a collaborative partnership will be developed between CHCs, health service research organizations, and academic researchers. The goal of the study is to examine the barriers that minority CHC patients face in receiving appropriate hypertension and diabetes care.

This study will develop a collaborative partnership between various health organizations and seven CHCs located in Boston neighborhoods that have a large percentage of African American and Hispanic residents. Researchers will conduct focus groups with CHC patients who are receiving care for hypertension or diabetes. CHC staff members will be interviewed to collect information regarding the relationship between CHC organizational structure and disparities in heart disease risk factors among minority patients with hypertension or diabetes. Researchers will then develop, implement, and evaluate a patient- and CHC-focused intervention aimed at reducing the cardiovascular risks of minority patients at four CHCs in Boston.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes
* Hypertension, as diagnosed by the average of two or more blood pressure measurements taken during two or more study visits following an initial screening
* Race is 'Black' or ethnicity is 'Hispanic'
* Patient at participating Community Health Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1204 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Potential outcomes for the future intervention include systolic blood pressure, diastolic blood pressure, and hemoglobin A1c | Measured from June to August 2008

CONTACTS AND LOCATIONS:
Overall Officials: LeRoi S. Hicks, MD, MPH, Principal Investigator — Harvard Medical School (HMS and HSDM); Thomas Keegan, PhD, Study Director — Harvard Medical School (HMS and HSDM)
Locations (2):
- United States (2):
  - Harvard Medical School, Boston, Massachusetts
  - Center for Community Health Education, Research, and Service, Boston, Massachusetts

REFERENCES:
- [Derived] Ndumele CD, Ableman G, Russell BE, Gurrola E, Hicks LS. Publication of recruitment methods in focus group research of minority populations with chronic disease: a systematic review. J Health Care Poor Underserved. 2011 Feb;22(1):5-23. doi: 10.1353/hpu.2011.0031. PMID 21317503
- [Derived] Russell BE, Gurrola E, Ndumele CD, Landon BE, O'Malley JA, Keegan T, Ayanian JZ, Hicks LS; Community Health and Academic Medicine Partnership Project. Perspectives of non-Hispanic Black and Latino patients in Boston's urban community health centers on their experiences with diabetes and hypertension. J Gen Intern Med. 2010 Jun;25(6):504-9. doi: 10.1007/s11606-010-1278-0. Epub 2010 Feb 24. PMID 20180156
- [Derived] Ndumele CD, Russell BE, Ayanian JZ, Landon BE, Keegan T, O'Malley AJ, Hicks LS. Strategies to improve chronic disease management in seven metro Boston community health centers. Prog Community Health Partnersh. 2009 Fall;3(3):203-11. doi: 10.1353/cpr.0.0080. PMID 19802379